CLINICAL TRIAL: NCT02029417
Title: OAG and Decitabine for Newly Diagnosed Acute Myeloid Leukemia Patients Greater Than or Equal to 65 Years of Age
Brief Title: Omacetaxine Mepesuccinate, Cytarabine, and Decitabine in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Major revisions needed in study
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 245213; NCI-2013-02425 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 245213 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Cytarabine; Homoharringtonine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cytarabine, omacetaxine mepesuccinate, decitabine) (Experimental): INDUCTION CHEMOTHERAPY: Patients receive cytarabine SC BID and omacetaxine mepesuccinate SC BID on days 1-14. Treatment for induction therapy repeats every 28 days for up to 4 courses or until patients achieve CR in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION THERAPY: Patients alternate courses between decitabine and OAG. Patients receive decitabine IV on days 1-5. Patients alternate with OAG courses, comprising cytarabine SC BID on days 1-7 and omacetaxine mepesuccinate SC BID on days 1-7. Treatment repeats every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cytarabine; Drug: omacetaxine mepesuccinate; Drug: decitabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cytarabine — Given SC
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: omacetaxine mepesuccinate — Given SC
  Other Names: CGX-635; homoharringtonine
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well omacetaxine mepesuccinate, cytarabine, and decitabine work in treating older patients with newly diagnosed acute myeloid leukemia. Omacetaxine mepesuccinate, cytarabine, and decitabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study the complete response rate following OAG (omacetaxine mepesuccinate, cytarabine) in newly diagnosed acute myeloid leukemia patients unfit for intensive induction therapy.

II. To assess the toxicity of OAG using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0).

SECONDARY OBJECTIVES:

I. To study the disease-free and overall survival of OAG and decitabine in newly diagnosed acute myeloid leukemia patients unfit for intensive induction therapy.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive cytarabine subcutaneously (SC) twice daily (BID) and omacetaxine mepesuccinate SC BID on days 1-14. Treatment for induction therapy repeats every 28 days for up to 4 courses or until patients achieve complete response (CR) in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY: Patients alternate courses between decitabine and OAG. Patients receive decitabine intravenously (IV) on days 1-5. Patients alternate with OAG courses, comprising cytarabine SC BID on days 1-7 and omacetaxine mepesuccinate SC BID on days 1-7. Treatment repeats every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not eligible for standard induction chemotherapy (or any standard therapy known to be life prolonging) because of poor performance status, significant tissue comorbidities, or unfavorable risk of disease
* Have an unequivocal histologic diagnosis of acute myeloid leukemia (AML) (including secondary AML)
* No prior therapy for AML except hydroxyurea to control counts
* Must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Subject or legal representative must understand the investigational nature of this study and sign an independent ethics committee/institutional review board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Subjects with the diagnosis of acute promyelocytic leukemia (t[15;17])
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the subject an unsuitable candidate to receive study drug
* Patients with sickle cell disease and sickle cell crisis
* Received an investigational agent for another disease within 30 days prior to enrollment
* The patient has an uncontrolled and active infection that would preclude study conduct and assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelena Ontiveros, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cytarabine, Omacetaxine Mepesuccinate, Decitabine): INDUCTION CHEMOTHERAPY: Patients receive cytarabine SC BID and omacetaxine mepesuccinate SC BID on days 1-14. Treatment for induction therapy repeats every 28 days for up to 4 courses or until patients achieve CR in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION THERAPY: Patients alternate courses between decitabine and OAG. Patients receive decitabine IV on days 1-5. Patients alternate with OAG courses, comprising cytarabine SC BID on days 1-7 and omacetaxine mepesuccinate SC BID on days 1-7. Treatment repeats every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  cytarabine: Given SC
  omacetaxine mepesuccinate: Given SC
  decitabine: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Cytarabine, Omacetaxine Mepesuccinate, Decitabine)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Cytarabine, Omacetaxine Mepesuccinate, Decitabine)
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of the Evaluable Population of Interest Who Experience a Complete Response in the Poor and Good Prognosis Groups
Description: Defined as recovery of morphologically normal bone marrow (< 5% blasts) and blood counts (absolute neutrophil count >= 1x10^9/L, platelet counts >= 100x10^9/LO) and rare circulating leukemic blasts or evidence of extramedullary disease. Analyzed using exact binomial probabilities in a two-stage design. The number of responses will be tabulated.
Time Frame: Up to 4 years
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Treatment (Cytarabine, Omacetaxine Mepesuccinate, Decitabine)
Number analyzed (Participants) | 0

2. Primary Outcome: Frequency of Adverse Events, Graded According to NCI CTCAE v4.0
Description: Maximum grade per participant of any AE.
Time Frame: Up to 30 days after last dose of study drugs
Population: All treated and eligible patients.
Measure: Number; unit: participants
Arm/Group | Treatment (Cytarabine, Omacetaxine Mepesuccinate, Decitabine)
Number analyzed (Participants) | 2
participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 2

ADVERSE EVENTS:
Arm/Group | Treatment (Cytarabine, Omacetaxine Mepesuccinate, Decitabine)
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cytarabine, Omacetaxine Mepesuccinate, Decitabine) (N=2)
Sepsis (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cytarabine, Omacetaxine Mepesuccinate, Decitabine) (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (4)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and low accrual no statistical inference of the primary aims were carried forth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes